CLINICAL TRIAL: NCT06854835
Title: The Value of Combined Detection of Different Blood Biomarkers in the Diagnosis and Treatments of Traumatic Brain Injury
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2020LSYY-G-269-01
Record Dates: First submitted 2025-01-06; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-01

CONDITIONS: Brain Injuries, Traumatic; Biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TBI, as a potential risk factor, causes a 1.5 times higher risk of neurodegenerative disease to up to 30-70% of TBI patients with neurological symptoms. Brain trauma is an important global medical, public health and social problem. Early diagnosis and effective treatment can effectively reduce the disability rate of patients and the incidence of neurological sequelae, and has increasingly become the focus of the international scientific research community. Exploring blood-based biomarkers has potential clinical value, which can greatly help clinicians to evaluate patients' conditions and develop reasonable plans, and then improve the clinical management and treatment of patients with craniocerebral trauma. Further research work is needed to be done to identify the most effective and efficient biomarker or combination marker strategies for integration into clinical treatment.

DETAILED DESCRIPTION:
Over the entire injury time phase of the TBI, the sampling of blood samples in the study was set within 24 hours, aiming to identify a set of biomarkers with assessment significance early after TBI. 1. The aim of this study was to investigate the correlation of different markers concentrations in blood and prognosis in patients with TBI. 2. Identify a set of biomarkers with assessment significance in the early period after TBI.

This project prospectively recruited 80 volunteer patients with voluntary TBI strictly in accordance with the inclusion and exclusion criteria, and 80 control groups matched by gender, age and education. 1 For patients who met the inclusion criteria, cranial MR and CT scans were performed at day 3 and discharge on admission, and clinical neuropsychological scale evaluation and peripheral whole blood collection were performed within 24 hours before each scan. 2. All fracture controls matched for sex, age, education and hands will complete primary MRI and CT examination, clinical neuropsychological scale evaluation and peripheral whole blood collection.Specific study contents include: 1. TBI patients were divided into mild, moderate and severe groups according to GCS scores, Together with the fracture patients in the control group, Blood and cerebrospinal fluid were collected from patients with TBI (mild: two blood collection after admission and discharge; Moderate and severe levels: admission, day 3, discharge, Take blood for three times and take cerebrospinal fluid once at admission); Blood of fracture patients (at admission) 2. Statistical analysis of clinical data. 3. Biomarker concentration determination: blood: NSE, GFAP, S100B, Tau, MBP (myelin basic protein), NFL; CSF: NSE, GFAP, Tau, NFL blood-brain barrier index (cerebrospinal fluid albumin / serum albumin). Among them, there was no dynamic monitoring, and comparison of blood and CSF markers in different groups. 4. Correlation analysis of blood markers, cerebrospinal fluid markers and the degree of brain injury (Spearman correlation analysis) shows the correlation between biomarkers and early assessment of the degree of TBI. 5. Follow-up was 3M / 6M, according to the GOS score: good prognosis and poor prognosis. 6. The correlation of serum and / or cerebrospinal fluid biomarker levels at admission and at discharge with GOS score (ROC curve).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old
2. Time of injury: patients with acute traumatic brain injury within 24h
3. Glasgow Coma Scale (Glasgow Coma Scale, GCS) score: 13 to 15 for patients with mild traumatic brain injury, 9 to 12 for moderate traumatic brain injury, and 3 to 8 for patients with severe traumatic brain injury
4. No other system damage has occurred
5. Admitted to hospital for the first diagnosis after the injury

Exclusion Criteria:

1. With a history of neurological or psychiatric disorders
2. Traumatic brain injury occurred before the injury
3. History of alcohol or substance abuse
4. Mild brain trauma is a complication of other injuries (systemic trauma, facial trauma, or spinal cord trauma) or other causes (psychological trauma, language impairment)
5. Patients without visits, and incomplete data during treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty voluntary TBI patients were recruited prospectively in strict accordance with the inclusion and exclusion criteria. Patients with TBI were divided into three groups: mild to moderate and severe according to GCS scores. At the same time, 80 limb fracture control group matched by gender, age and education were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Full Outline of Unresponsiveness, FOUR | On admission (within 24 hours), 3 days of admission and at discharge (up to 24 weeks)
  The FOUR is an questionnaire which has four main assessments: eye opening, exercise, brain stem reflex, and respiratory function. Each item has a full score of 4 and a total score of 16. Brainstem reflex and respiratory function of FOUR are more sensitive than the GCS language score for predicting mortality risk in ICU patients. The total score was 0 to 16, with lower scores indicating a greater probability of death and disability.
Glasgow Outcome Scale-Extended, GOS-E | On admission (within 24 hours), 3 days of admission and at discharge (up to 24 weeks)
  GOS-E is a clinical assessment tool for assessing function and quality of life in patients with head trauma. This is an expanded version of the Glasgow Rating Scale, designed to provide a more comprehensive assessment to better understand the patient's recovery. The GOS-E scores were divided into the following categories: 1= death, 2= vegetative state, 3= severe disability, 4= moderate to severe disability, 5= moderate disability, 6= mild disability, 7= good recovery, and 8= complete recovery
Head MRI | On admission (within 24 hours), 3 days of admission and at discharge (up to 24 weeks)
  The MRI scan sequence includes the following:
  1. 3-pl (positioning image requires preservation of the whole brain, including overhead scalp to all cerebellum) (check the parameters before scanning)
  2. T2-FLAIR (predict brain conditions, if abnormal lesions, stop scanning immediately)
  3. ESWAN
  4. T1-weighted 3D-MPRAGE
  5. DTI
  6. Resting State (BOLD) (positioning line is parallel to AC-PC line)
  7. ASL
  8. Axial-T1

IPD SHARING:
Plan to Share IPD: No